CLINICAL TRIAL: NCT06506942
Title: The TRICURE EFS TRiCares Topaz Transfemoral TRICUspid Heart Valve REplacement System Early Feasibility Study
Brief Title: The TRICURE EFS Study
Acronym: TRICURE EFS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TRiCares (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2301
Record Dates: First submitted 2024-07-11; First posted 2024-07-18 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Tricuspid Valve Regurgitation; Heart Valve Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Heart Valve Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transcatheter Tricuspid Valve Replacement (Experimental): Treatment with the TRiCares Topaz Tricuspid Transcatheter Valve Replacement System
  Interventions: Device: Transcatheter Tricuspid Valve Replacement

INTERVENTIONS:
Device: Transcatheter Tricuspid Valve Replacement — Replacement of the tricuspid valve through a transcatheter approach
  Other Names: TRiCares Topaz Tricuspid Valve Replacement System

SUMMARY:
Prospective, multi-center study to assess safety and performance of the TRiCares Topaz Tricuspid Valve Replacement System

DETAILED DESCRIPTION:
The study is a multi-center, prospective single arm study designed to evaluate the safety and performance of the TRiCares Topaz Tricuspid Valve Replacement System.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Tricuspid regurgitation grade 3 (severe) on a scale of 0 (none) to 5 (torrential)
* Institutional Heart Team evaluates patient as being at increased operative risk

Exclusion Criteria:

* Patient in need of emergent intervention
* Patient who is hemodynamically unstable
* Anatomical contraindications for implantation with study device
* Patient who is currently participating in another clinical investigation where the primary endpoint was not reached yet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Composite of MAE | 30 day post-intervention
  Composite rate of major adverse events (MAEs) at 30 days, including mortality, myocardial infarction, stroke and major complications.
Device Success | immediately post-intervention
  Device success defined as a reduction in tricuspid regurgitation immediately post-intervention

SECONDARY OUTCOMES:
Six minute walk test | 30 days, 6 months, annual for five years post-intervention
  Change in distance (m) compared to baseline assessment
Reduction in Tricuspid Regurgitation (TR) Grade | 30 days, 6 months, annual for five years post-intervention
  Number of patients presenting with reduction in TR grade compared to baseline assessment
New York Heart Association (NYHA) Function Class | 30 days, 6 months, annual for five years post-intervention
  Number of patients presenting with improvement in NYHA classification

CONTACTS AND LOCATIONS:
Overall Officials: Susheel Kodali, MD, Principal Investigator — Columbia University Medical Center/ NewYork Presbyterian Hospital; Gorav Ailawadi, MD, Principal Investigator — University of Michigan Hospital and Health Systems
Locations (8):
- United States (8):
  - Piedmont Healthcare Inc., Atlanta, Georgia
  - Northwestern, Chicago, Illinois
  - University of Michigan Hospital and Health Systems, Ann Arbor, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Columbia University Medical Center/ NewYork Presbyterian Hospital, New York, New York
  - Montefiore, The Bronx, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No